CLINICAL TRIAL: NCT00003989
Title: Phase II Trial With ISIS 3521/CGP 64128A in Patients With Malignant Melanoma and Non Small Cell Lung Cancer
Brief Title: ISIS 3521 in Treating Patients With Advanced, Unresectable, or Metastatic Non-small Cell Lung Cancer or Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16977; EORTC-16977; ISIS-EORTC-16977
Record Dates: First submitted 1999-11-01; First posted 2004-08-27 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer; Melanoma (Skin)
Keywords: recurrent non-small cell lung cancer; stage III melanoma; stage IV melanoma; recurrent melanoma; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — ISIS 3521

INTERVENTIONS:
Biological: ISIS 3521

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ISIS 3521 in treating patients who have advanced, unresectable, or metastatic non-small cell lung cancer or unresectable or metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete and partial response rates and duration of response in patients with locally advanced, unresectable, or metastatic non-small cell lung cancer or unresectable or metastatic melanoma treated with ISIS 3521. II. Determine safety of ISIS 3521 in these patients.

OUTLINE: This is a multicenter study. Patients are stratified by disease type. Patients receive ISIS 3521 IV over 21 days followed by 7 days of rest. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 28-50 patients (14-25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven melanoma that is unresectable and regionally metastatic, or widely disseminated OR Histologically or cytologically proven non-small cell lung cancer (NSCLC) that is locally advanced, unresectable, or metastatic Stage IIIA, IIIB, or IV Evidence of disease progression prior to study At least 1 bidimensionally measurable lesion The following are NOT considered measurable: previously irradiated lesions, ascites, pleural effusion, bone metastases, brain metastases, leptomeningeal disease, or an abdominal mass that can be palpated but not measured Melanoma patients whose only manifestation of disease is 1 of the following are NOT eligible: Lymphedema Pleural effusion Ascites CNS metastases Bone marrow infiltration Osteoblastic bone lesions

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 No abnormal clotting tests Hepatic: Bilirubin no greater than 2.0 mg/dL AST and ALT no greater than 2 times upper limit of normal (ULN) (5 times ULN if due to liver metastases) Renal: Creatinine no greater than 1.6 mg/dL OR Creatinine clearance at least 60 mL/min Urinary protein less than 0.3 g/dL Cardiovascular: No superior vena cava obstruction in NSCLC unless successfully treated at least 2 months prior to study Other: No underlying disease state associated with active bleeding No prior or concurrent malignancies at other sites except adequately treated cone biopsied carcinoma in situ of the cervix uteri or basal cell or squamous cell skin cancer No nonmalignant systemic disease making patient poor risk for study No active uncontrolled infection Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy (including interferon or interleukin-2) for melanoma patients No other concurrent anticancer immunotherapy Chemotherapy: No prior chemotherapy for melanoma patients except adjuvant or local chemotherapy (extracorporeal circulation) At least 4 weeks since prior adjuvant or local chemotherapy if presence of measurable lesions outside the treated limb (6 months if no presence of measurable lesions outside the treated limb) No prior chemotherapy for NSCLC except platinum compounds used as radiosensitizer At least 4 weeks since prior platinum compounds No other concurrent anticancer chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Concurrent radiotherapy allowed for bone pain or other reasons No irradiation of all evaluable lesions Surgery: See Disease Characteristics Other: At least 4 weeks since other prior investigational drugs No other concurrent investigational drugs No concurrent anticoagulants except heparin used to prevent occlusion of IV lines during week(s) off treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Shoshana Kaplan, MD, Study Chair — Universitaetsspital-Basel
Locations (27):
- Austria (2):
  - Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna (Wien)
- Belgium (4):
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Ludwig Institute for Cancer Research-Brussels Branch, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Herlev, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Universitaetsklinik und Strahlenklinik - Essen, Essen
  - Klinikum Nurnberg, Nuremberg (Nurnberg)
- Netherlands (5):
  - Academisch Ziekenhuis der Vrije Universiteit, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - St. Radboud University Hospital, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - Saint Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - C.R.C. Beatson Laboratories, Glasgow, Scotland